CLINICAL TRIAL: NCT06876818
Title: Predictive Cardio-Metabolic Trascrictomics Trajectories in the Barilla Offspring Follow-Up STUDY: the PREDICT-OMICS Study.
Brief Title: Predictive Cardio-Metabolic Trascrictomics Trajectories in the Barilla Offspring Follow-Up Study
Acronym: PREDICT-OMICS
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: University of Parma (Other)
Responsible Party: Principal Investigator, Alessandra Dei Cas, Prof., Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: 604-2023; 2022FZL247 (Other Grant/Funding Number: PRIN-2022)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer
Keywords: transcriptomic analysis; cardio-metabolic analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — PBMC, monocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants in the Barilla Offspring Study
  Interventions: Other: Evaluation of transcriptomic and cardio-metabolic profiles

INTERVENTIONS:
Other: Evaluation of transcriptomic and cardio-metabolic profiles — The parameters and variables collected in 2006-2007 (T0) will be re-evaluated at the follow-up visit (T1), including demographic, anthropometric, lifestyle data (smoking habit, physical activity, sleep quality) blood pressure, standard biochemical analysis and inflammatory profile. To assess the evolution of glucose tolerance and vascular damage, metabolic (OGTT) and cardiovascular (carotid ecodoppler) profile analyses will be repeated. For gene expression analyses, in addition to messenger RNA from PBMCs (as at T0), RNA from PBMC-derived monocytes will also be extracted and sequenced at T1.

SUMMARY:
Experimental, drug-free, longitudinal, single-centre study for the prediction of cardiometabolic risk in Barilla Off-Spring Study subjects by analysing the evolution of transcriptomic signatures

DETAILED DESCRIPTION:
In Westernized societies, common metabolic and cardiovascular diseases have complex etiologies involving dynamic genome-metagenome-environment interactions. The early molecular alterations that initiate and sustain their progression, although still only partially understood, are thought to share common roots in the terrain of insulin resistance (IR). In recent decades, reciprocal relationships between IR and inflammation have been unraveled, leading to the general concept of "meta-inflammation". In turn, the regulatory role played by metabolic signatures in immune cells has led to the concept of "immunometabolism". In particular, in these meta-inflammation-related disorders, there is a paucity of prospective gene expression data, especially in the early stages of their natural history. Gene expression profiling of peripheral blood mononuclear cells (PBMCs) may be a useful and accessible window into the pathophysiology of processes occurring in difficult-to-access organs and tissues. In a deeply phenotyped healthy cohort, the Barilla Offspring Study, a transcriptomic signature exclusively associated with IR was found by analyzing PBMC gene expression with a novel rank-based classification method, which was also found to discriminate diseased from healthy individuals in Alzheimer's disease, chronic heart failure and type 2 diabetes. The granularity of this approach can be further improved by examining gene expression in monocytes, as cells of innate immunity and mainly implicated in inflammatory/degenerative disorders and their risk factors. In this longitudinal study, we aim to identify the transcriptomic signature(s) in circulating immune cells and inflammatory biomarkers that predict or are associated with 15-year changes in glucose tolerance and/or carotid artery atherogenic phenotype. The study has solid premises: i. The cohort of subjects offers a unique opportunity to identify PBMC transcriptomic trajectories (baseline and 15-year follow-up) that predict changes in cardiometabolic phenotype; ii. cross-sectional assessment of monocyte transcriptomic profiling in the same cohort may uncover additional lineage-specific signatures associated with different cardio-metabotypes at follow-up, allowing comparison with PBMC; iii. an innovative rank-based classification method - SCUDO and its extensions - will be used, in addition to standard methods, to compute transcriptomic analyses. The results of the study may identify cellular transcriptomic signatures and trajectories, which could link cardiometabolic phenotypes at the molecular and cellular level, highlighting possible biological mechanisms of cardiometabolic disease susceptibility and progression, and unveiling a wide range of molecular targets in PBMC and, especially, monocytes, which can be further investigated for their validity as peripheral biomarkers for risk assessment. The findings will also provide new insights into targeted pharmacological strategies for the prevention and/or treatment of cardiometabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the Barilla Off-Spring Study (2006-2007)
* Ability to understand the methods, aims and implications of the study, and to give free and informed consent

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults who participated in the cross-sectional Barilla Offspring Study in 2006-2007
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Selection of a set of candidate genes directly correlated with the development of altered metabolic phenotypes | within six months of the enrolment visit
  All data related to the transcriptomics of PBMCs at T0 (2006-2007) will be retrieved. At T1, a blood sample will be collected from which PBMCs will be isolated. Total RNA will be purified and its quality tested using the Quibit fluorimetric technique and the Tape-station system. From the same blood sample, the monocyte subpopulation will also be isolated and used to identify the specific transcriptomic signature.
  Both RNA datasets, collected at T0 and T1, will be processed to identify informative transcriptomic signatures of baseline and follow-up conditions. The sets will be converted to obtain a profile for a symbol gene; this will allow easier comparison of the calculated transcriptomic signatures between different datasets, facilitating the biological interpretation of the results.

SECONDARY OUTCOMES:
Selection of a set of candidate genes directly related to the development of altered vascular phenotypes | within six months of the enrolment visit
  All data related to the transcriptomics of PBMCs at T0 (2006-2007) will be retrieved. At T1, a blood sample will be collected from which PBMCs will be isolated. Total RNA will be purified and its quality tested using the Quibit fluorimetric technique and the Tape-station system. From the same blood sample, the monocyte subpopulation will also be isolated and used to identify the specific transcriptomic signature.
  Both RNA datasets, collected at T0 and T1, will be processed to identify informative transcriptomic signatures of baseline and follow-up conditions. The sets will be converted to obtain a profile for a symbol gene; this will allow easier comparison of the calculated transcriptomic signatures between different datasets, facilitating the biological interpretation of the results.
Selection of a set of candidate genes directly related to overt altered metabolic and/or vascular phenotypes. | within six months of the enrolment visit
  All data related to the transcriptomics of PBMCs at T0 (2006-2007) will be retrieved. At T1, a blood sample will be collected from which PBMCs will be isolated. Total RNA will be purified and its quality tested using the Quibit fluorimetric technique and the Tape-station system. From the same blood sample, the monocyte subpopulation will also be isolated and used to identify the specific transcriptomic signature.
  Both RNA datasets, collected at T0 and T1, will be processed to identify informative transcriptomic signatures of baseline and follow-up conditions. The sets will be converted to obtain a profile for a symbol gene; this will allow easier comparison of the calculated transcriptomic signatures between different datasets, facilitating the biological interpretation of the results.
Selection of markers directly related to the development of altered metabolic and/or vascular phenotypes. | within six months of the enrolment visit
  All data related to the transcriptomics of PBMCs at T0 (2006-2007) will be retrieved. At T1, a blood sample will be collected from which PBMCs will be isolated. Total RNA will be purified and its quality tested using the Quibit fluorimetric technique and the Tape-station system. From the same blood sample, the monocyte subpopulation will also be isolated and used to identify the specific transcriptomic signature.
  Both RNA datasets, collected at T0 and T1, will be processed to identify informative transcriptomic signatures of baseline and follow-up conditions. The sets will be converted to obtain a profile for a symbol gene; this will allow easier comparison of the calculated transcriptomic signatures between different datasets, facilitating the biological interpretation of the results.
Selection of a set of candidate genes directly related to alterations in biohumoral parameters and the inflammatory profile. | within six months of the enrolment visit
  All data related to the transcriptomics of PBMCs at T0 (2006-2007) will be retrieved. At T1, a blood sample will be collected from which PBMCs will be isolated. Total RNA will be purified and its quality tested using the Quibit fluorimetric technique and the Tape-station system. From the same blood sample, the monocyte subpopulation will also be isolated and used to identify the specific transcriptomic signature.
  Both RNA datasets, collected at T0 and T1, will be processed to identify informative transcriptomic signatures of baseline and follow-up conditions. The sets will be converted to obtain a profile for a symbol gene; this will allow easier comparison of the calculated transcriptomic signatures between different datasets, facilitating the biological interpretation of the results.
Selection of a set of candidate genes directly related to alterations in lifestyle. | within six months of the enrolment visit
  All data related to the transcriptomics of PBMCs at T0 (2006-2007) will be retrieved. At T1, a blood sample will be collected from which PBMCs will be isolated. Total RNA will be purified and its quality tested using the Quibit fluorimetric technique and the Tape-station system. From the same blood sample, the monocyte subpopulation will also be isolated and used to identify the specific transcriptomic signature.
  Both RNA datasets, collected at T0 and T1, will be processed to identify informative transcriptomic signatures of baseline and follow-up conditions. The sets will be converted to obtain a profile for a symbol gene; this will allow easier comparison of the calculated transcriptomic signatures between different datasets, facilitating the biological interpretation of the results.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Department of Medicine and Surgery, Parma, PR, Italy

REFERENCES:
- [Background] Scazzina F, Dei Cas A, Del Rio D, Brighenti F, Bonadonna RC. The beta-cell burden index of food: A proposal. Nutr Metab Cardiovasc Dis. 2016 Oct;26(10):872-8. doi: 10.1016/j.numecd.2016.04.015. Epub 2016 May 6. PMID 27381989
- [Background] Bianchi C, Miccoli R, Trombetta M, Giorgino F, Frontoni S, Faloia E, Marchesini G, Dolci MA, Cavalot F, Cavallo G, Leonetti F, Bonadonna RC, Del Prato S; GENFIEV Investigators. Elevated 1-hour postload plasma glucose levels identify subjects with normal glucose tolerance but impaired beta-cell function, insulin resistance, and worse cardiovascular risk profile: the GENFIEV study. J Clin Endocrinol Metab. 2013 May;98(5):2100-5. doi: 10.1210/jc.2012-3971. Epub 2013 Mar 28. PMID 23539736
- [Background] Myhrstad MC, Ulven SM, Gunther CC, Ottestad I, Holden M, Ryeng E, Borge GI, Kohler A, Bronner KW, Thoresen M, Holven KB. Fish oil supplementation induces expression of genes related to cell cycle, endoplasmic reticulum stress and apoptosis in peripheral blood mononuclear cells: a transcriptomic approach. J Intern Med. 2014 Nov;276(5):498-511. doi: 10.1111/joim.12217. Epub 2014 Mar 20. PMID 24641624
- [Background] Chi H. Immunometabolism at the intersection of metabolic signaling, cell fate, and systems immunology. Cell Mol Immunol. 2022 Mar;19(3):299-302. doi: 10.1038/s41423-022-00840-x. Epub 2022 Feb 21. No abstract available. PMID 35190684
- [Background] Ahlqvist E, Storm P, Karajamaki A, Martinell M, Dorkhan M, Carlsson A, Vikman P, Prasad RB, Aly DM, Almgren P, Wessman Y, Shaat N, Spegel P, Mulder H, Lindholm E, Melander O, Hansson O, Malmqvist U, Lernmark A, Lahti K, Forsen T, Tuomi T, Rosengren AH, Groop L. Novel subgroups of adult-onset diabetes and their association with outcomes: a data-driven cluster analysis of six variables. Lancet Diabetes Endocrinol. 2018 May;6(5):361-369. doi: 10.1016/S2213-8587(18)30051-2. Epub 2018 Mar 5. PMID 29503172
- [Background] Adeva-Andany MM, Martinez-Rodriguez J, Gonzalez-Lucan M, Fernandez-Fernandez C, Castro-Quintela E. Insulin resistance is a cardiovascular risk factor in humans. Diabetes Metab Syndr. 2019 Mar-Apr;13(2):1449-1455. doi: 10.1016/j.dsx.2019.02.023. Epub 2019 Feb 22. PMID 31336505